CLINICAL TRIAL: NCT00672971
Title: An Open Label Randomized Study to Compare the Safety and Efficacy of Silcap Plus (Approximately 4% Dimeticone) Against Nix Cream Rinse.
Brief Title: Safety and Efficacy Study to Compare a 4% Dimethicone Foam and Nix Cream Rinse (1% Permethrin) in the Control of Head Lice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Bart Rossel, Managing Director, Oystershell NV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OYS001-07
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Head Lice
MeSH Terms: interventions — Permethrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 4% dimethicone foam
  Interventions: Other: 4% dimethicone foam
- 2 (Active Comparator): 1% permethrin
  Interventions: Other: 1% permethrin

INTERVENTIONS:
Other: 4% dimethicone foam — The dimethicone foam is applied to dry hair and left on the hair for approximately 15 minutes. The product is then removed by washing the hair with baby shampoo. The foam is applied two time, separated by an interval of 7-9 days.
  Other Names: Oxykal, Neo-paraderma
  Arms: 1
Other: 1% permethrin — Nix® Cream Rinse is applied as indicated on the product labeling. The cream rinse is applied to wet hair and left on the hair for 10 minutes. The hair is then rinsed with tepid water to remove the product, toweled dry, and combed with a detangling comb. The product is applied two times, separated by an interval of 7-9 days.
  Other Names: Nix cream rinse
  Arms: 2

SUMMARY:
The purpose of this study was to evaluate the efficacy of a dimethicone foam in the control of head lice and to compare the efficacy to a permethrin based product.

ELIGIBILITY:
Inclusion Criteria:

* 4 - 85 years of age
* active head lice infestation of at least ≥ 10 live lice
* short hair (hair no longer than 2 inches below the neck) or long hair (hair 2 inches below the neck to mid back)

Exclusion Criteria:

* had received or used an investigational new drug within the 30 days immediately preceding the study
* used any form of head lice treatment whether prescription, over-the-counter, or a home remedy for at least fourteen days prior to their study visit
* used topical medication of any kind on the hair for a period of 48 hours prior to the visit
* had a history of allergy to rag weed, permethrin, or mineral oil, or had taken trimethoprim or cotrimoxazole at evaluation or during the previous four weeks
* Female subjects that were pregnant or breast feeding

Ages: 4 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Cure rate at the final visit (Day 14 or 15). Cure rate was defined as the number of subjects free of live head lice divided by the total number of subjects in the treatment group (x 100). | 14 or 15 days after 1st treatment

SECONDARY OUTCOMES:
Any adverse events during or after application of the product | up to 7 or 8 d after product application

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Serrano, CRI, Principal Investigator — Lice Source Services
Locations (1):
- Lice Source Services Inc, Plantation, Florida, United States